CLINICAL TRIAL: NCT01947088
Title: I. The Effect of Music Therapy on Cognitive Recovery From Pediatric Epilepsy Surgery
Brief Title: Effect of Music Therapy on Cognitive Recovery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left facility
Sponsor: Seton Healthcare Family (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CR-13-087
Record Dates: First submitted 2013-08-27; First posted 2013-09-20 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Epilepsy
Keywords: Epilepsy, seizure disorder
MeSH Terms: conditions — Epilepsy | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Therapy Arm (Experimental): Music therapy evaluation prior to surgery (Baseline 1). These evaluations will also be given within 3 days of epilepsy surgery (Baseline 2), 8 weeks after surgery (Baseline 3), and 9-12 months after surgery (Baseline 4.) Pre-study and post-study scores from the neuropsychological assessments will be compared to determine if music therapy has a significant effect on the child's cognitive recovery. Will consist of meeting with the music therapists, Certified Child Life Specialists (CCLS), or Child Life Assistants (CLA) for music therapy (treatment group) for about 45 minutes, twice per week, for Weeks 1-8. CThe Music Therapy group will partake in interventions such as singing and playing musical instruments.
  Interventions: Behavioral: Music Therapy
- Unstructured Play Arm (Active Comparator): Child life programs provide children with opportunities to engage in normal play and recreational activities that promote growth, development and feelings of success and fulfillment.All brain surgery candidates receive a neuropsychological assessment before and after surgery (9-12 months after surgery). This is the standard of care for all brain surgery patients. The results of this assessment and will be used in this research study. In addition, patients who agree to participate in the study will receive cognitive screening and a music therapy evaluation prior to surgery (Baseline 1). These evaluations will also be given within 3 days of epilepsy surgery (Baseline 2), 8 weeks after surgery (Baseline 3), and 9-12 months after surgery (Baseline 4.)
  Interventions: Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — Will consist of meeting with the music therapists, Certified Child Life Specialists (CCLS), or Child Life Assistants (CLA) for either music therapy for about 45 minutes, twice per week, for Weeks 1-8. The Music Therapy group will partake in interventions such as singing and playing musical instruments. All brain surgery candidates receive a neuropsychological assessment before and after surgery (9-12 months after surgery). In addition, patients who agree to participate in the study will receive cognitive screening and a music therapy evaluation prior to surgery (Baseline 1). These evaluations will also be given within 3 days of epilepsy surgery (Baseline 2), 8 weeks after surgery (Baseline 3), and 9-12 months after surgery (Baseline 4.)

SUMMARY:
Participation in music therapy will result in improvement in cognitive functioning, as measured by neuropsychological testing 9-12 months following surgery.

DETAILED DESCRIPTION:
Music therapy could have a significant impact on clinical outcomes for patients with epilepsy. One study found that epilepsy patients who received music therapy for six months or greater had a significant reduction in number of seizures and could potentially aid in decreasing medication dosage. The investigators would like to contribute to this sort of research, but focus on what effect music therapy has on a patient's cognitive recovery after undergoing epilepsy surgery. Although research exists regarding music therapy on memory and communication, its overall effect on this patient population is unclear.

The Dell Children's Epilepsy program hopes that this research project on memory and communication will have a positive effect on their patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Between 6-16 years of age
* Will undergo either a brain resection or lobectomy

Exclusion Criteria:

* Pre-surgical Full Scale IQ below 70
* Primary language is not English
* Hearing or vision impairments
* Parental consent cannot be obtained

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Participation in music therapy will result in improvement in neuropsychological scores 12 months following surgery for music therapy study group. | 12 months post surgery
  All brain surgery candidates receive a neuropsychological assessment before and after surgery (9-12 months after surgery). This is the standard of care for all brain surgery patients. The results of this assessment and will be used in this research study. In addition, patients who agree to participate in the study will receive cognitive screening and a music therapy evaluation prior to surgery (Baseline 1). These evaluations will also be given within 3 days of epilepsy surgery (Baseline 2), 8 weeks after surgery (Baseline 3), and 9-12 months after surgery (Baseline 4.)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Townsend, MMT, Principal Investigator — Seton Healthcare Family
Locations (1):
- Dell Children's Medical Center of Central Texas, Austin, Texas, United States